CLINICAL TRIAL: NCT02223520
Title: Treating Parents to Reduce Neonatal Intensive Care Unit (NICU) Transmission of Staphylococcus Aureus
Brief Title: Treating Parents to Reduce NICU Transmission of Staphylococcus Aureus Trial
Acronym: TREAT PARENTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NA_00092982; R01HS022872 (AHRQ)
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2020-03

CONDITIONS: Staph Aureus Colonization; Staph Aureus Infection
Keywords: Staphylococcus aureus; Infection; Colonization; Transmission; Neonate
MeSH Terms: conditions — Staphylococcal Infections; Infections | interventions — Mupirocin; Chlorhexidine; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mupirocin and Chlorhexidine (Active Comparator): Participants will apply 2% intranasal mupirocin twice a day for five days and cleanse with 2% chlorhexidine cloths once a day for five days.
  Interventions: Drug: Mupirocin and Chlorhexidine
- Placebo ointment and placebo cloths (Placebo Comparator): Participants will apply 2% petrolatum intranasal placebo ointment twice a day for five days and cleanse with 2% non-medicated soap placebo cloths once a day for five days.
  Interventions: Drug: Placebo ointment and placebo cloths

INTERVENTIONS:
Drug: Mupirocin and Chlorhexidine
  Other Names: bactroban; chlorhexidine gluconate
  Arms: Mupirocin and Chlorhexidine
Drug: Placebo ointment and placebo cloths
  Arms: Placebo ointment and placebo cloths

SUMMARY:
This trial will test the hypothesis that treating parents of neonates requiring NICU care with intranasal mupirocin and topical chlorhexidine bathing will reduce the spread of S. aureus from parents to neonates.

DETAILED DESCRIPTION:
The TREAT PARENTS Trial, or Treating Parents to Reduce NICU Transmission of S. aureus, is a placebo-controlled, double-masked, randomized clinical trial to test the hypothesis that treatment of S. aureus colonized parents with intranasal mupirocin and topical chlorhexidine gluconate antisepsis will decrease neonatal S. aureus acquisition. All neonates admitted to the Johns Hopkins Hospital and Johns Hopkins Bayview Medical Center NICUs will be pre-screened and parents will be approached for enrollment in the study. After consent and baseline screening, 400 neonate-parent pairs will be randomized; only neonates who have a parent colonized with S. aureus will be randomized. Parents will receive a 5 day treatment with intranasal mupirocin plus topical chlorhexidine gluconate antisepsis or placebo.

After recruitment and informed consent, parents will undergo pre-randomization screening. If both parents screen negative for S. aureus colonization, the neonate will be ineligible for the randomization and parents will be informed that the parents are not colonized at that time with S. aureus. If either parent screens positive for S. aureus, then both parents as a pair will be eligible for randomization to one of the two possible masked treatment arms. The neonate-parent "pair" will be the unit of randomization and each parent will be allocated to the same group if both consent.

After the baseline neonate testing for S. aureus colonization, repeat testing will be performed every 7 days for the neonates until the neonate acquires S. aureus colonization or is discharged from the NICU.

ELIGIBILITY:
Inclusion Criteria:

* Neonate has never had a clinical or surveillance culture grow S. aureus
* Neonate was transferred from another hospital or admitted from home and had admission screening cultures for S. aureus colonization that were negative (if admission cultures were not performed, the cultures will be performed as part of the pre-randomization screening process)
* Parent(s) is(are) able to visit the child at the bedside
* Parent(s) test positive for S. aureus at screening
* Neonate has anticipated stay longer than 5 days in the NICU (if estimated stay is unclear, parents can be screened for S. aureus colonization and decision to randomize can be delayed until hospital day 3 or 4 after reassessment of anticipated stay).
* Parents is(are) willing to be randomized
* No documented or reported allergies to any agent used in either treatment regimen
* Able to perform written informed consent

Exclusion Criteria:

* Allergies to any agent used in either treatment regimen
* Neonate has had a prior clinical or surveillance culture grow S. aureus
* Neonate admitted to NICU from home and is greater than 7 days of age
* Neonate admitted to NICU from another hospital and is greater than 7 days of age
* Neonate is a ward of the State
* Not able to provide written informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Milstone, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland

REFERENCES:
- [Derived] Milstone AM, Voskertchian A, Koontz DW, Khamash DF, Ross T, Aucott SW, Gilmore MM, Cosgrove SE, Carroll KC, Colantuoni E. Effect of Treating Parents Colonized With Staphylococcus aureus on Transmission to Neonates in the Intensive Care Unit: A Randomized Clinical Trial. JAMA. 2020 Jan 28;323(4):319-328. doi: 10.1001/jama.2019.20785. PMID 31886828
- [Derived] Milstone AM, Koontz DW, Voskertchian A, Popoola VO, Harrelson K, Ross T, Aucott SW, Gilmore MM, Carroll KC, Colantuoni E. Treating Parents to Reduce NICU Transmission of Staphylococcus aureus (TREAT PARENTS) trial: protocol of a multisite randomised, double-blind, placebo-controlled trial. BMJ Open. 2015 Sep 9;5(9):e009274. doi: 10.1136/bmjopen-2015-009274. PMID 26353875

RESULTS

PARTICIPANT FLOW:
Groups:
- Mupirocin and Chlorhexidine: Participants will apply 2% intranasal mupirocin twice a day for five days and cleanse with 2% chlorhexidine cloths once a day for five days.
  Mupirocin and Chlorhexidine
- Placebo Ointment and Placebo Cloths: Participants will apply 2% petrolatum intranasal placebo ointment twice a day for five days and cleanse with 2% non-medicated soap placebo cloths once a day for five days.
  Placebo ointment and placebo cloths
Period: Overall Study
Arm/Group | Mupirocin and Chlorhexidine | Placebo Ointment and Placebo Cloths
Started | 147 | 160
Completed | 147 (101 neonates of these parents were enrolled. 12 were lost to follow-up.) | 160 (107 neonates of these parents were enrolled. 6 were lost to follow-up.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mupirocin and Chlorhexidine | Placebo Ointment and Placebo Cloths | Total
Number analyzed (Participants) | 147 | 160 | 307
Age, Continuous [Mean (Standard Deviation); unit: days] — Age of neonate at time of enrollment (days) Population: This baseline measure reported is for the neonates not the parents.
  days
    number analyzed (Participants) | 101 | 107 | 208
    (all) | 7.9 (5.1) | 7.2 (5.3) | 7.54 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This baseline measure reported is for the neonates not the parents.
  Participants
    number analyzed (Participants) | 101 | 107 | 208
    Female | 47 | 47 | 94
    Male | 54 | 60 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: This baseline measure reported is for the neonates not the parents.
  Participants
    number analyzed (Participants) | 101 | 107 | 208
    Hispanic or Latino | 8 | 3 | 11
    Not Hispanic or Latino | 86 | 95 | 181
    Unknown or Not Reported | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: This baseline measure reported is for the neonates not the parents.
  Participants
    number analyzed (Participants) | 101 | 107 | 208
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 3 | 11 | 14
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 27 | 30 | 57
    White | 66 | 59 | 125
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 5 | 7 | 12
Region of Enrollment [Count of Participants; unit: Participants] — Population: This baseline measure reported is for the neonates not the parents.
  Participants
    United States: number analyzed (Participants) | 101 | 107 | 208
    United States: Johns Hopkins Hospital | 93 | 99 | 192
    United States: Johns Hopkins Bayview | 8 | 8 | 16
Parent age at the time of enrollment [Mean (Standard Deviation); unit: years] — Population: This is a measure for the parents. Parent demographics collected by parent interview or parent completion of form. Parents sometimes skipped questions on survey form and were not always available to capture missing demographic data that was not in the medical record.
  years
    number analyzed (Participants) | 134 | 146 | 280
    (all) | 30.3 (5.9) | 30.9 (7.7) | 30.6 (6.9)
Parent antibiotic use in past 6 months [Count of Participants; unit: Participants]
  Yes | 59 | 54 | 113
  No | 73 | 88 | 161
  Unreported/Unknown | 15 | 18 | 33
Parent history of mupirocin use [Count of Participants; unit: Participants]
  Yes | 6 | 5 | 11
  No | 121 | 133 | 254
  Unreported/Unknown | 20 | 22 | 42
Parent history of Staphylococcus aureus infection [Count of Participants; unit: Participants]
  Yes | 6 | 9 | 15
  No | 122 | 128 | 250
  Unreported/Unknown | 19 | 23 | 42
Level of education of parent [Count of Participants; unit: Participants]
  At most high school | 26 | 33 | 59
  Some or completed college | 71 | 59 | 130
  Graduate degree | 24 | 38 | 62
  Unknown | 26 | 30 | 56
No. of singletons [Count of Participants; unit: Participants] — Neonates that were delivered as singletons. Population: This baseline measure reported is for the neonates not the parents.
  Participants
    number analyzed (Participants) | 101 | 107 | 208
    (all) | 78 | 81 | 159
Birthweight of neonate [Mean (Standard Deviation); unit: grams] — Population: This baseline measure reported is for the neonates not the parents.
  grams
    number analyzed (Participants) | 101 | 107 | 208
    (all) | 1982.5 (972.8) | 1986.9 (949.4) | 1984.8 (958.5)
Child delivery method [Count of Participants; unit: Participants] — Population: This baseline measure reported is for the neonates not the parents.
  Participants
    number analyzed (Participants) | 101 | 107 | 208
    Vaginal birth | 68 | 72 | 140
    Cesarean section | 33 | 35 | 68
Neonate inborn or transferred in [Count of Participants; unit: Participants] — Inborn was defined as neonates who were born at Johns Hopkins Hospital (JHH)/Johns Hopkins Bayview Medical Center (JHBMC) instead of being transferred to JHH/JHBMC from an outside hospital or home. Population: This baseline measure reported is for the neonates not the parents.
  Participants
    number analyzed (Participants) | 101 | 107 | 208
    Inborn in JHH/JHBMC | 91 | 97 | 188
    Transferred from another hospital to JHH/JHBMC | 10 | 8 | 18
    Transferred from home to JHH/JHBMC | 0 | 2 | 2
Gestational age at birth [Mean (Standard Deviation); unit: weeks] — Population: This baseline measure reported is for the neonates not the parents.
  weeks
    number analyzed (Participants) | 101 | 107 | 208
    (all) | 32.9 (4.7) | 33.1 (4.4) | 33 (4.5)
Maternal antibiotic use during delivery [Count of Participants; unit: Participants] — Neonates whose mothers reported using antibiotic during delivery. Population: This baseline measure reported is for the neonates not the parents.
  Participants
    number analyzed (Participants) | 101 | 107 | 208
    (all) | 68 | 64 | 132
Maternal Group B Streptococcus positive [Count of Participants; unit: Participants] — Neonates whose mothers reported testing positive for Group B Streptococcus. Population: This baseline measure reported is for the neonates not the parents.
  Participants
    number analyzed (Participants) | 101 | 107 | 208
    Positive | 21 | 21 | 42
    Negative | 32 | 43 | 75
    Unreported/Unknown | 48 | 43 | 91
Maternal HIV Positive [Count of Participants; unit: Participants] — Neonates whose mothers reported being positive for HIV. Population: This baseline measure reported is for the neonates not the parents.
  Participants
    number analyzed (Participants) | 101 | 107 | 208
    Positive | 1 | 2 | 3
    Negative | 92 | 94 | 186
    Unreported/Unknown | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Neonatal Infections With a S. Aureus Strain That is Concordant to Parental S. Aureus Strain
Description: Primary outcome is neonatal acquisition of S. aureus strain that is concordant to parental S. aureus strain as determined by periodic surveillance cultures or a culture collected during routine clinical care that grows S. aureus. Survival analysis techniques will be used to compare the hazard of concordant colonization comparing Treatment and Control Groups.
Time Frame: Up to 90 days
Population: This outcome is being assessed in the neonate population not the mothers. 12 of the neonates in the intervention group and 6 in the placebo group were lost to follow-up and could not be included in the analysis.
Measure: Number; unit: neonatal S. aureus infections
Arm/Group | Mupirocin and Chlorhexidine | Placebo Ointment and Placebo Cloths
Number analyzed (Participants) | 89 | 101
neonatal S. aureus infections | 13 | 29

ADVERSE EVENTS:
Time Frame: During the 5 days of treatment
Description: Adverse events were assessed in mothers not neonates.
Arm/Group | Mupirocin and Chlorhexidine | Placebo Ointment and Placebo Cloths
All-Cause Mortality (participants affected / at risk) | 0/147 | 0/160
Serious Adverse Events (participants affected / at risk) | 0/147 | 0/160
Other Adverse Events (participants affected / at risk) | 9/147 | 16/160
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mupirocin and Chlorhexidine (N=147) | Placebo Ointment and Placebo Cloths (N=160)
Skin irritation (Skin and subcutaneous tissue disorders) | 7 (7) | 10 (10)
Nose irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Retained placenta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT02223520/Prot_SAP_000.pdf